CLINICAL TRIAL: NCT02641054
Title: Double-Blind Randomized Placebo-Controlled Cross-Over Phase IIa Trial to Evaluate Efficacy of CVXL-0107 on Parkinson-Related Symptoms and Levodopa-Induced Dyskinesia in Advanced Parkinson's Disease Patients Using a Levodopa Challenge Test
Brief Title: Efficacy Phase IIa Study of CVXL-0107 in Advanced Parkinson's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CleveXel Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CT-CVXL-0107-01
Record Dates: First submitted 2015-12-07; First posted 2015-12-29 (Estimated); Last update posted 2017-07-24 (Actual); Status verified 2017-07

CONDITIONS: Idiopathic Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Levodopa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CVXL-0107 then cross-over to placebo (Experimental): Study drug (CVXL-0107) 4 times per day for 2 weeks on top of usual treatment for Parkinson disease, followed by one challenge test day: one intake of study drug on top of supraoptimal dose of levodopa.
  Cross-over to placebo 4 times per day for 2 weeks on top of usual treatment for Parkinson disease, followed by one challenge test day: one intake of placebo on top of supraoptimal dose of levodopa
  Interventions: Drug: CVXL-0107; Drug: Placebo; Drug: Levodopa
- Placebo then cross-over to CVXL-0107 (Placebo Comparator): Placebo 4 times per day for 2 weeks on top of usual treatment for Parkinson disease, followed by one challenge test day: one intake of placebo on top of supraoptimal dose of levodopa.
  Cross-over to study drug (CVXL-0107) 4 times per day for 2 weeks on top of usual treatment for Parkinson disease, followed by one challenge test day: one intake of study drug on top of supraoptimal dose of levodopa
  Interventions: Drug: CVXL-0107; Drug: Placebo; Drug: Levodopa

INTERVENTIONS:
Drug: CVXL-0107
Drug: Placebo
Drug: Levodopa

SUMMARY:
CVXL-0107 a glutamate release inhibitor, has shown evidence of antiparkinsonian and antidyskinetic activity in a macaque model and has shown a significant effect on the UPDRS-III (Movement Disorder Society - Unified Parkinson's Disease Rating Scale) while "ON", as well as an increase of "ON-time" without dyskinesia or without troublesome dyskinesia in a previous phase 2a proof of concept study. This study will confirm the efficacy of CVXL-0107 in combination with optimal dose of levodopa on motor symptoms of Parkinson's disease (PD) .

DETAILED DESCRIPTION:
Phase IIa study, 1:1 randomized, double blind placebo- controlled, with cross-over. Each volunteer patient will be randomly assigned to receive CVXL-0107 or placebo as add-on PD therapy and crossed-over to the other arm in the second sequence of the study. They will be assessed during an acute levodopa challenge test with one intake of the study drug or placebo with a supra-optimal dose of levodopa after 2 weeks of daily treatment with the same study drug or placebo. Patients will be cross-overed to the other treatment and reassessed during a second acute levodopa challenge test after 2 weeks of daily treatment with the study drug or the placebo. The study will evaluate the anti-PD and the anti-dyskinesia efficacy of CVXL-0107 as measured by MDS-UPDRS part III (Movement Disorder Society - Unified Parkinson's Disease Rating Scale) and on levodopa-induced dyskinesia as measured by the AIMS (Abnormal Involuntary Movement Scale).

ELIGIBILITY:
Inclusion Criteria:

1. Signed written Informed Consent
2. Male and female patient aged 40 -75 years
3. Clinical diagnosis of idiopathic PD according to the UK Parkinson's Disease Society Brain Bank Clinical Diagnosis Criteria
4. Advanced PD with clear daily motor fluctuations and dyskinesia with optimal levodopa-based therapy
5. At least 2 hours in "OFF" state per day including morning OFF
6. Predictable "OFF" in the morning on awakening prior to receiving morning dose of levodopa
7. During an acute levodopa challenge test : Motor improvement of at least 30% on the MDS-UPDRS part III and AIMS score ≥ 1 at least two time points
8. Patient with dyskinesia: MDS-UPDRS items 4.1 ("time spent with dyskinesia") and 4.2 ("functional impact of dyskinesia") scores ≥ 1 at Screening
9. Hoehn and Yahr stages of 2-4 in the "OFF" state at Screening
10. Stable doses and regimens of antiparkinsonian medications for at least the last month prior to randomization (levodopa, dopamine agonists and selective monoamine oxidase type B inhibitors (selegiline, rasagiline))
11. Anti-PD therapy intended to remain constant throughout the course of the study
12. Normal platelets count
13. Mini-mental state examination (MMSE)≥24 at Screening
14. PD patient treated by DBS can be included if surgery occurred at least one year before the study
15. Patient with health insurance
16. Female of childbearing potential with an effective contraception

Exclusion Criteria:

1. Any relevant neurologic or psychiatric disease, except idiopathic PD
2. Any secondary causes for Parkinsonism or other neurodegenerative disorder with Parkinsonism symptoms
3. Any neurosurgical intervention for PD planned during the study period
4. Neuroleptics and any D2-receptor antagonists within the last 3 months before Screening
5. Amantadine, Riluzole, dextromethorphan, apomorphine continuous infusion (pump), morphine, or memantine, during the last month before screening and during the study duration
6. History of psychosis or treatment with any antipsychotic drugs within the last 2 years
7. History of seizure or epilepsy, or treatment with anticonvulsant drugs within the last year
8. Any clinically significant unstable medical illness in the last month before randomization (e.g. unstable angina, unstable vascular disease etc)
9. Anti-cancer treatment within the 3 months before Screening
10. Treatment with anticoagulant drugs
11. Any clinically significant renal (serum creatinine level ≥1.5x ULN or dialysis) or hepatic (liver enzyme values≥2x ULN) disease
12. Any clinically significant condition that may compromise the safety of patient or the conduct of the study protocol according to Investigators' opinion.
13. Known genetic disorder of human UDP-glucuronosyltransferase
14. Participation in another trial with any investigational product within the last month before randomization or intake of any investigational product
15. Pregnant, breastfeeding or lactating female

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Change in MDS-UPDRS part III (Movement Disorder Society - Unified Parkinson's Disease Rating Scale Part III) score. | at visit 3 (day 15= challenge test day) and visit 4 (day 37= challenge test day): at baseline (before L-Dopa administration), then every 20 minutes during the first hour and then every 30 minutes during 5 hours.
  CVXL-0107 and placebo
Change in AIMS ( Abnormal Involuntary Movement Scale) score | at visit 3 (day 15= challenge test day) and visit 4 (day 37 = challenge test day): at baseline (before L-Dopa administration), then every 20 minutes during the first hour and then every 30 minutes during 5 hours
  CVXL-0107 and placebo

SECONDARY OUTCOMES:
Incidence of Clinical Treatment-Emergent Adverse Events [Safety and Tolerability] | at visit 3 (day 14) and visit 4 (day 36)
  Physical examination, vital signs
Hematology laboratory safety of CVXL-0107 | at visit 3 (day 14) and visit 4 (day 36)
  complete blood count
Hepatic laboratory safety of CVXL-0107 | at visit 3 (day 14) and visit 4 (day 36)
  aspartate transaminase, alanine transaminase, gamma-glutamyl-transpeptidase, alkaline phosphatase
Area Under the Curve [AUC] of CVXL-0107 concentrations | at visit 3 (day 15= challenge test day) and visit 4 (day 37= challenge test day)
  Blood samples at L-dopa intake and after 20', 40', 60', 90', 120', 240'.
Area Under the Curve [AUC] of levodopa concentrations | at visit 3 (day 15= challenge test day) and visit 4 (day 37= challenge test day)
  Blood samples at L-dopa intake and after 20', 40', 60', 90', 120', 240'.
Assessment of total daily "ON" time in Patients Diaries | During 3 days, prior to visit 3 (days 11-13) and prior to visit 4 (days 33, 34, 35)
  Total "ON-time"
Assessment of daily "ON" time without dyskinesia in Patients Diaries | During 3 days; prior to visit 3 (days 11-13) and prior to visit 4 (days 33, 34, 35)
  "ON-time" without dyskinesia

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Christophe Corvol, MD, PhD, Principal Investigator — CIC-Neurologie, bâtiment ICM, Hôpital Pitié-Salpêtrière, 47/83 Bd de l'Hôpital, 75013 Paris, France
Locations (1):
- Clevexel Pharma, Maisons-Alfort, France

IPD SHARING:
Plan to Share IPD: No